CLINICAL TRIAL: NCT01792024
Title: Phase II Evaluation of MR-Guided Laser Induced Interstitial Thermal Therapy (LITT) for Prostate Cancer
Brief Title: MR-Guided Laser Interstitial Thermal Therapy in Treating Patients With Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-1841; NCI-2013-00404 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R21CA173751 (NIH)
Record Dates: First submitted 2013-02-12; First posted 2013-02-15 (Estimated); Results first posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-02

CONDITIONS: Stage I Prostate Cancer; Stage II Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (LITT) (Experimental): Patients undergo Magnetic Resonance imaging (MR) guided laser thermal therapy with Visualase Thermal Therapy device.
  Interventions: Device: Visualase Thermal Therapy; Procedure: magnetic resonance imaging

INTERVENTIONS:
Device: Visualase Thermal Therapy — MR guided laser ablation of prostate cancer
  Other Names: laser interstitial thermal therapy
Procedure: magnetic resonance imaging — Undergo MR-guided LITT
  Other Names: MRI; NMR imaging; NMRI; nuclear magnetic resonance imaging

SUMMARY:
This phase II trial studies how well magnetic resonance (MR)-guided laser interstitial thermal therapy works in treating patients with prostate cancer. Laser therapy uses intense, narrow beams of light to cut and destroy tissue and may help treat prostate cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the oncologic efficacy of laster interstitial thermal therapy (LITT) with primary endpoint of undetectable cancer on magnetic resonance imaging (MRI)-guided biopsy of treatment zone at 3 months following treatment.

SECONDARY OBJECTIVES:

I. To evaluate oncologic efficacy at 12 months following treatment based on biopsy of the treatment zone.

II. To determine treatment-related safety and toxicity. III. To longitudinally assess urinary and sexual function in the year following treatment.

OUTLINE:

Patients undergo MR-guided LITT.

After completion of study treatment, patients are followed up at 1, 3, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Clinical characteristics:

  * Stage T1c or T2a
  * Prostate-specific antigen (PSA) < 15 ng/ml or PSA density (PSA divided by prostate volume in cubic centimeters) < 0.15 ng/ml^3
* No evidence of metastatic disease based on National Comprehensive Cancer Network (NCCN) guidelines:

  * Bone scan if PSA > 20 ng/ml and clinical stage T1c
  * Bone scan if PSA > 10 ng/ml and clinical stage T2
* Biopsy requirements:

  * Gleason score 7 or less
  * 25% or fewer biopsies with cancer
  * At least 12 biopsy cores of the prostate
  * Within 12 months of treatment
* Imaging requirements:

  * Up to 2 visible magnetic resonance (MR) lesion(s) concordant with sextant of biopsy-detected cancer(s)
  * MRI within 6 months of treatment
* Karnofsky performance status of at least 70
* General health is suitable to undergo the planned minimally invasive procedures
* Risks, benefits, and alternatives discussed with informed consent given

Exclusion Criteria:

* Previous treatment of prostate cancer with luteinizing hormone releasing hormone (LHRH) agonist/antagonist, chemotherapy, surgery, or radiation
* Presence of 3 or more visible lesions on MRI
* High suspicion of seminal vesicle invasion or lymph node metastases on MRI
* Unable to tolerate MRI (medical device, foreign body, claustrophobia, body habitus, or other)
* Renal insufficiency with estimated glomerular filtration rate (eGFR) < 30 ml/min/body surface area (BSA) based on Modification in Diet Renal Disease equation; inability to safely receive gadolinium contrast for MRI
* History of prior pelvic surgery with surgical clips remaining in situ (e.g., bladder, bowel, internal pelvic organs) that compromise MRI image quality
* Other serious illnesses involving the cardiac, respiratory, central nervous system (CNS), or hepatic organ systems, which would preclude study completion or impede the determination of causality of any complications experienced during the conduct of this study

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-01-28 (Actual); Primary Completion 2015-09-16 (Actual); Study Completion 2015-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aytekin Oto, Principal Investigator — University of Chicago Comprehensive Cancer Center; Scott Eggener, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (LITT): Patients undergo MR-guided laser ablation of prostate cancer
  Visualase Thermal Therapy: MR guided laser ablation of prostate cancer
  magnetic resonance imaging: Undergo MR-guided LITT
Period: Overall Study
Arm/Group | Treatment (LITT)
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (LITT)
Number analyzed (Participants) | 27
Age, Continuous [Median (Full Range); unit: years] | 62 [47 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Undetectable Cancer on MRI-guided Biopsy of Ablation Zone Following Treatment
Description: The primary study end point was the number of patients with no cancer on MRI guided biopsy of the ablation zone at 3 months.
Time Frame: At 3 months after ablation
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (LITT)
Number analyzed (Participants) | 27
Participants | 26

2. Secondary Outcome: The Number of Patients With Biopsy Cancer of the Treatment Zone
Description: A systematic 12-core biopsy was performed at 1 year and the number of patients with biopsy cancer was counted.
Time Frame: At 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (LITT)
Number analyzed (Participants) | 27
Participants | 3

3. Secondary Outcome: The Total Number of Patients With Any Adverse Events Related to the Treatment
Description: Treatment-related toxicity measured by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.0
Time Frame: 1,3, and 12 month after treatment and up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (LITT)
Number analyzed (Participants) | 27
Participants | 20

4. Secondary Outcome: Quality of Life in Terms of Urinary and Sexual Function in the Year Following Treatment Assessed Using the International Prostate Symptom Score (IPSS)
Description: International Prostate Symptom Score (IPSS) measures urinary symptoms and continence and it ranged 0 to 35. Lower values are considered better outcome.
Time Frame: At 1,3 and 12 months
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Treatment (LITT)
Number analyzed (Participants) | 27
units on a scale
  At 1 month | 10 [1 to 21]
  At 3 month | 7 [0 to 25]
  At 12 month | 10 [1 to 26]

5. Secondary Outcome: Quality of Life in Terms of Urinary and Sexual Function in the Year Following Treatment Assessed Using Sexual Health Inventory in Men (SHIM)
Description: Sexual Health Inventory Score in Men (SHIM) measures sexual health and erectile function and it ranged 1 to 25. Lower values are considered better outcome.
Time Frame: At 1,3 and 12 months
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Treatment (LITT)
Number analyzed (Participants) | 27
units on a scale
  At 1 month | 19 [1 to 25]
  At 3 month | 19 [1 to 25]
  At 12 month | 21 [3 to 25]

ADVERSE EVENTS:
Time Frame: 1,3 and 12 months after treatment
Arm/Group | Treatment (LITT)
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 2/27
Other Adverse Events (participants affected / at risk) | 20/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (LITT) (N=27)
Bleeding per rectum (Injury, poisoning and procedural complications) | 1
Fever (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (LITT) (N=27)
Allergic reaction (Immune system disorders) | 2
Erectile dysfunction (Reproductive system and breast disorders) | 5
Hematuria (Renal and urinary disorders) | 9
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 3
Scrotal pain (Reproductive system and breast disorders) | 2
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 6
Urinary frequency (Renal and urinary disorders) | 2
urinary incontinence (Renal and urinary disorders) | 2
Urinary retention (Renal and urinary disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No